CLINICAL TRIAL: NCT01293513
Title: Structured Treatment Interruption (STI) in Acute/Primary HIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof. Israel Yust, Kobler AIDS Center, Tel Sourasky Medical Center ISRAEL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-10-IY-0190-10-TLV-CTIL
Record Dates: First submitted 2011-02-08; First posted 2011-02-10 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2011-02

CONDITIONS: HIV Infections
Keywords: Only patients with Acute or Primary HIV infection will be studied
MeSH Terms: conditions — HIV Infections | interventions — Treatment Interruption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Gradual anti-HIV treatment interruption — Gradual interruption of anti-HIV treatment: the interruption initially for a week, up to six weeks' interruption, and continuing anti-HIV treatment for two weeks between successive interruptions
  Other Names: STI (Structured treatment interruption)

SUMMARY:
Although the introduction of Highly Active Anti-Retroviral Therapy - HAART - has dramatically altered the course of HIV/AIDS, true cure is still unattainable and patients are required to take these medications for the rest of their lives. As is well known, the prolonged use of such agents is associated with serious, sometimes life-threatening side effects, metabolic disturbances such as diabetes and an increased incidence of myocardial infarction.

In 1999, a patient with acute HIV infection was treated soon after diagnosis ("Berlin patient"). However because of intercurrent conditions, treatment was interrupted on two occasions. After the third introduction of therapy, treatment was terminated (arbitrarily) and the patient was found to have undetectable virus throughout a follow up of approximately 18 months. The possible explanation of this phenomenon was autovaccination. Other workers have tried Structured Treatment Interruption (STI) in Acute/Primary HIV Infection with controversial results, possibly because there were too few cycles of treatment interruption.

In a patient treated in our center for Acute HIV infection, after initial HAART therapy, he underwent gradually increasing interruptions of treatment from 1 to 7 weeks. After complete cessation of treatment, the patient was followed for 3 years, where CD4 levels were normal, CD4/CD8 ratio remained above 1 and the viral load was undetectable.

Our plan is to study patients with Acute/Primary HIV Infection, who have been treated with HAART for at least one year. Once they have been shown to have undetectable virus (less than 40 copies HIV RNA per milliliter) and CD4 above 500 per microliter with a CD4/CD8 above 1, they can be enrolled in the STI study.

The study will comprise 6 groups of 4 cycles of treatment/interruption with an increasing duration treatment interruptions alternating with treatment intervals over a 33 month period. Altogether there will be 24 treatment interruptions, lasting from 1 week to 6 weeks. During this time the patients will be regularly monitored for clinical events and laboratory parameters.

The purpose of the study is to determine whether patients with acute/primary HIV infection undergoing graded STI can achieve a normal immune status and undetectable viral load on a long-term basis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Acute HIV infection, where the time from infection to seroconversion is from 6 to 12 weeks
* Patients with Primary HIV infection, where the time from appearance of HIV antibodies seroconversion until the setpoint is less than 6 months
* Post menopausal females or potentially fertile women who agree either to refrain from sexual relations or to use contraceptive devices
* Patients who are willing to participate and who understand the trial, can read and sign the agreement form prior to entering the study

Exclusion Criteria:

* Patients suffering from serious disease, including hepatic or renal insufficiency and following organ transplantation
* Pregnant females or potentially fertile women who are unwilling to refrain from sexual relations or to use contraceptive devices
* Patients requiring chemotherapy or radiotherapy up till six months before entering the trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
CD4 Cells normal value and Viral load undetectable (<50 per ml) | 33 months